CLINICAL TRIAL: NCT06566989
Title: An Open-label Phase 1 Study to Evaluate Metabolism, Excretion, and Mass Balance of [¹⁴C]MK-5684 in Healthy Male Participants
Brief Title: A Study of the Absorption, Distribution, Metabolism, and Elimination of Opevesostat (MK-5684) in Healthy Adult Male Participants (MK-5684-008)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Collaborators: Orion Corporation, Orion Pharma (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 5684-008; MK-5684-008 (Other: MSD); 1010197 (Registry Identifier: IRAS)
Record Dates: First submitted 2024-08-20; First posted 2024-08-22 (Actual); Last update posted 2024-10-23 (Actual); Status verified 2024-10

CONDITIONS: Metastatic Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Prednisone; Fludrocortisone; fludrocortisone acetate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- [¹⁴C]Opevesostat (Experimental): On Day 1, participants receive a single dose of [¹⁴C]opevesostat as an oral solution. Participants then receive single doses of 5.0 mg prednisone and 0.05 mg fludrocortisone tablets 4 hours later as hormone replacement therapy.
  Interventions: Drug: [¹⁴C]Opevesostat; Drug: Prednisone; Drug: Fludrocortisone

INTERVENTIONS:
Drug: [¹⁴C]Opevesostat — Oral solution
  Other Names: MK-5684
Drug: Prednisone — Tablet
  Other Names: RAYOS®; STERAPRED®; DELTASONE®
Drug: Fludrocortisone — Tablet
  Other Names: FLORINEF®

SUMMARY:
This is a study of opevesostat in healthy adult male participants. The purpose of this study is to understand the absorption, distribution, metabolism, and elimination of opevesostat in humans, as well as its pharmacokinetics (PK), metabolic profile, and safety and tolerability.

ELIGIBILITY:
Inclusion Criteria:

* Is a healthy male according to the assessment of the investigator
* Has a body mass index of 18.0 to 32.0 kg/m2
* Has regular bowel movements (i.e., average stool production of ≥1 and ≤3 stools per day)

Exclusion Criteria:

* Has the presence or history of clinically significant allergy requiring treatment
* Has a history of adrenal insufficiency
* Has veins not suitable for multiple venipunctures/cannulation
* Has previously taken part in more than 3 radiolabeled drug studies in the last 12 months
* Has donated blood or plasma within the previous 3 months or lost greater than 400 mL of blood

Ages: 30 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 8 (Actual)
Dates: Start 2024-09-19 (Actual); Primary Completion 2024-10-17 (Actual); Study Completion 2024-10-17 (Actual)

PRIMARY OUTCOMES:
Cumulative amount of total radioactivity excreted in urine (CumAeu) after administration of single-dose [¹⁴C]Opevesostat | Predose and at designated time points (up to 8 days)
  Urine samples will be collected at pre-specified timepoints and used to determine CumAeu.
Cumulative amount of total radioactivity excreted in feces (CumAef) after administration of single-dose [¹⁴C]Opevesostat | Predose and at designated time points (up to 8 days)
  Fecal samples will be collected at pre-specified timepoints and used to determine CumAef.
Cumulative percentage of total radioactivity excreted in urine (Cumfeu) after administration of single-dose [¹⁴C]Opevesostat | Predose and at designated time points (up to 8 days)
  Urine samples will be collected at pre-specified timepoints and used to determine CumFeu.
Cumulative percentage of total radioactivity excreted in feces (Cumfef) after administration of single-dose [¹⁴C]Opevesostat | Predose and at designated time points (up to 8 days)
  Fecal samples will be collected at pre-specified timepoints and used to determine Cumfef.
Plasma Opevesostat Pharmacokinetics: Area under the curve from time 0 to the time of last measurable concentration (AUC0-t) | Predose and at designated time points (up to 8 days)
  Plasma samples will be collected at pre-specified timepoints and used to determine AUC0-t of opevesostat.
Plasma Opevesostat Pharmacokinetics: Area under the curve from time 0 to extrapolated infinity (AUC0-inf) | Predose and at designated time points (up to 8 days)
  Plasma samples will be collected at pre-specified timepoints and used to determine AUC0-inf of opevesostat.
Plasma Opevesostat Pharmacokinetics: Maximum observed concentration (Cmax) | Predose and at designated time points (up to 8 days)
  Plasma samples will be collected at pre-specified timepoints and used to determine Cmax of opevesostat.
Plasma Opevesostat Pharmacokinetics: Time of maximum observed concentration (Tmax) | Predose and at designated time points (up to 8 days)
  Plasma samples will be collected at pre-specified timepoints and used to determine Tmax of opevesostat.
Plasma Opevesostat Pharmacokinetics: Terminal elimination half-life (t1/2) | Predose and at designated time points (up to 8 days)
  Plasma samples will be collected at pre-specified timepoints and used to determine t1/2 of opevesostat.
Plasma Total Radioactivity Pharmacokinetics: Area under the curve from time 0 to the time of last measurable concentration (AUC0-t) | Predose and at designated time points (up to 8 days)
  Plasma samples will be collected at pre-specified timepoints and used to determine AUC0-t of total radioactivity.
Plasma Total Radioactivity Pharmacokinetics: Area under the curve from time 0 to extrapolated infinity (AUC0-inf) | Predose and at designated time points (up to 8 days)
  Plasma samples will be collected at pre-specified timepoints and used to determine AUC0-inf of total radioactivity.
Plasma Total Radioactivity Pharmacokinetics: Maximum observed concentration (Cmax) | Predose and at designated time points (up to 8 days)
  Plasma samples will be collected at pre-specified timepoints and used to determine Cmax of total radioactivity.
Plasma Total Radioactivity Pharmacokinetics: Time of maximum observed concentration (Tmax) | Predose and at designated time points (up to 8 days)
  Plasma samples will be collected at pre-specified timepoints and used to determine Tmax of total radioactivity.
Plasma Total Radioactivity Pharmacokinetics: Terminal elimination half-life (t1/2) | Predose and at designated time points (up to 8 days)
  Plasma samples will be collected at pre-specified timepoints and used to determine t1/2 of total radioactivity.
Total Number of Metabolites in Plasma that Represent at least 10% of the Dose of Radioactivity | Predose and at designated time points (up to 8 days)
  Plasma samples will be collected at pre-specified timepoints and used to determine the total number of metabolites that represent at least 10% of the dose of radioactivity. Metabolites will be determined using liquid scintillation and high-resolution mass spectrometry.
Total Number of Metabolites in Urine that Represent at least 10% of the Dose of Radioactivity | Predose and at designated time points (up to 8 days)
  Urine samples will be collected at pre-specified timepoints and used to determine the total number of metabolites that represent at least 10% of the dose of radioactivity. Metabolites will be determined using liquid scintillation and high-resolution mass spectrometry.
Total Number of Metabolites in Feces that Represent at least 10% of the Dose of Radioactivity | Predose and at designated time points (up to 8 days)
  Fecal samples will be collected at pre-specified timepoints and used to determine the total number of metabolites that represent at least 10% of the dose of radioactivity. Metabolites will be determined using liquid scintillation and high-resolution mass spectrometry.

SECONDARY OUTCOMES:
Number of Participants with One or More Adverse Events (AEs) | Up to approximately 8 days
  An AE is any untoward medical occurrence in a clinical study participant, temporally associated with the use of study intervention, whether or not considered related to the study intervention. An AE can therefore be any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease (new or exacerbated) temporally associated with the use of study intervention. The number of participants who experienced an AE will be reported.
Number of Participants who Discontinue from the Study Due to an AE | Up to approximately 8 days
  An AE is any untoward medical occurrence in a clinical study participant, temporally associated with the use of study intervention, whether or not considered related to the study intervention. An AE can therefore be any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease (new or exacerbated) temporally associated with the use of study intervention. The number of participants who discontinue from the study due to an AE will be reported.

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC
Locations (1):
- Quotient Sciences ( Site 0001), Nottingham, Nottinghamshire, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
http://engagezone.msd.com/doc/ProcedureAccessClinicalTrialData.pdf
URL: http://engagezone.msd.com/ds_documentation.php

REFERENCES:
- See also: Merck Clinical Trials Information — https://www.merckclinicaltrials.com/